CLINICAL TRIAL: NCT01977378
Title: A Double-Blind,Venlafaxine-Controlled Study of Efficacy and Safety of Sustained-Release Desvenlafaxine Hydrochloride in the Treatment of Major Depressive Disorder
Brief Title: A Study of Sustained-Release Desvenlafaxine Hydrochloride for the Treatment of Major Depressive Disorder
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DVS20130806
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-10

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sustained-Release Desvenlafaxine Hydrochloride (Experimental): 50-100mg/d
  Interventions: Drug: Sustained-Release Desvenlafaxine Hydrochloride
- Sustained-Release Venlafaxine Hydrochloride (Active Comparator): 75-225mg/d
  Interventions: Drug: Sustained-Release Venlafaxine Hydrochloride

INTERVENTIONS:
Drug: Sustained-Release Desvenlafaxine Hydrochloride
  Arms: Sustained-Release Desvenlafaxine Hydrochloride
Drug: Sustained-Release Venlafaxine Hydrochloride
  Arms: Sustained-Release Venlafaxine Hydrochloride

SUMMARY:
A multicenter, 10-week study to evaluate the efficacy and safety of Sustained-Release Desvenlafaxine Hydrochloride versus Sustained-Release venlafaxine Hydrochloride in adult with major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Adult with primary diagnosis of Major Depressive Disorder
* Aged from 18 years to 65 years
* A primary diagnosis of Major Depressive Disorder based on the criteria in the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM- IV-TR), single or recurrent episode, without psychotic features
* Hamilton Psychiatric Rating Scale for Depression (HAM-D 17) total score of ≧ 20
* Clinical Global Impressions Scale-Severity (CGI-S) score of ≧4

Exclusion Criteria:

* Known hypersensitivity to desvenlafaxine or venlafaxine
* Significant risk of suicide based on clinical judgment
* Women who were pregnant,breast-feeding,or planning to become pregnant during study
* Had a history of seizure disorder
* History or current evidence of gastrointestinal disease known to interfere with the absorption or excretion of drugs or a history of surgery known to interfere with the absorption or excretion of drugs
* Any unstable hepatic, renal, pulmonary, cardiovascular, ophthalmologic, neurologic, or other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results
* Cancer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline on the Hamilton Rating Scale for Depression, 17-item Total Score (HAM-D17) | Baseline to Week 10

SECONDARY OUTCOMES:
Change From Baseline on the Clinical Global Impression Scale | Baseline to Week 10
Change From Baseline in Clinical Global Impression-Improvement (CGI-I) Scale | Baseline to Week 10
Change From Baseline in Sheehan Disability Scale (SDS) Total Score at Week 10 | Baseline to Week 10
Change From Baseline in Adjusted Mean on Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline to Week 10
Change From Baseline on the Visual Analogue Scale-Pain Intensity (VAS-PI) | Baseline to Week 10
Number of Participants in Remission Based on the HAM-D17 at Week 10 | Baseline to Week 10
  Remission was defined as a HAM-D17 score of less than or equal to 7.

CONTACTS AND LOCATIONS:
Overall Officials: Huafang Li, Professor, Principal Investigator — The Shanghai Mental Health
Locations (6):
- China (6):
  - Guangdong General Hospital, Guangzhou, Guangdong
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - West China Hospital, Chengdu, Sichuan
  - Beijing An Ding Hospital, Beijing
  - Beijing HuiLongGuan Hospital, Beijing
  - The Shanghai Mental Health, Shanghai